CLINICAL TRIAL: NCT06204250
Title: A Phase 1 Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of GS1-144 Tablets
Brief Title: A Study to Assess Safety and Tolerability of GS1-144 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: GenSci074-102
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Vasomotor Symptoms; Adult Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 Single Ascending Dose: Cohorts 1 to 6 (Experimental): Participants will receive GS1-144 5 mg, 15 mg, 30 mg, 60 mg , 90 mg and 120mg tablets once on Day 1 in their respective Cohort in Part 1. 2 participants will receive placebo in each cohort.
  Interventions: Drug: GS1-144; Drug: Placebo
- Part 2 Multiple Ascending Dose: Cohorts 1 to 4 (Experimental): tablets once on Day 1 in their respective Cohort in Part 2. 2 participants will receive placebo in each cohort.
  Interventions: Drug: GS1-144; Drug: Placebo

INTERVENTIONS:
Drug: GS1-144 — Oral tablets.
Drug: Placebo — Matching placebo tablets.

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of single ascending doses of GS1-144 in healthy participants in Part 1 and to assess the safety and tolerability of multiple ascending doses of GS1-144 in healthy postmenopausal female participants in Part 2.

DETAILED DESCRIPTION:
This study will be divided into two sequential parts: Part 1 single ascending dose (SAD), and Part 2 multiple ascending dose (MAD) with the overall design.

Part 1 will enroll a total of approximately 46 healthy participants in five cohorts at 5 milligram (mg), 15 mg, 30 mg, 60 mg and 90 mg dose levels. Each cohort will have 2 participants receiving placebo. There is no restriction on the male-to female ratio.

Part 2 will be conducted after confirming the safety and tolerability of the ->30mg dose in Part 1 and will enroll a total of approximately 30 healthy postmenopausal female participants and provisionally consists of three cohorts at 15 mg, 30 mg 60 mg and 120mg dose levels. Each cohort will have 2 participants receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form (ICF): Part 1 only: healthy male and female participants aged between 18 and 45 years inclusive; Part 2 only: healthy women aged between 40 and 65 years inclusive who have undergone natural menopause;
2. Body weight >=50 kilogram (kg) (male), >=45 kg (female) with a body mass index between 18.0 and 32.0 kilogram per square meter (kg/m^2) inclusive at screening;
3. Part 1 only: Female participants are eligible to participate if they are not pregnant, not breastfeeding, and highly effective contraception includes placement of an intrauterine device or intrauterine system plus use of a condom;
4. Part 1 only: Male participants must agree to practice true abstinence; be surgically sterilized; or agree to use a condom plus effective contraception for their female partner, if of childbearing potential, from screening and for at least 90 days after dosing and refrain from donating sperm during this period. These contraception requirements do not apply if the male participant is in an exclusively same sex relationship;
5. Able to comprehend the nature of the study and any risks associated with participation and willing to cooperate and comply with protocol restrictions and requirements.

Exclusion Criteria:

1. Any known allergy to the components or analogues of the investigational product, or those with an allergic constitution;
2. A history of currently suffering from any other cardiovascular, gastrointestinal, endocrine, hematological, hepatic, immunological, metabolic, urinary, pulmonary, neurological, dermatological, psychiatric, renal and/or other major diseases deemed clinically significant by the investigator;
3. Known/confirmed history of malignancy;
4. A history of epileptic seizure or increased risk of epileptic seizure, or participants with a recent history of head trauma leading to loss of consciousness or concussion;
5. A history of currently suffering from hypothalamic dysfunction;
6. Significant acute/chronic infections within two weeks prior to dosing;
7. Undergone major surgical procedures within six months prior to screening or plan to undergo any surgery during the trial;
8. Participated in other clinical trials within 1 month prior to dosing;
9. Have lost or donated more than 400 mL of blood within 1 month prior to screening;
10. Have taken any prescription/over-the-counter drugs or dietary supplements within 7 days prior to dosing or within 5 halflives of the drug;
11. Clinically significant abnormalities on physical examination or genitourinary ultrasound at the time of screening;
12. Clinically significant abnormalities in vital signs;
13. Prolonged QTcF interval in 12-lead ECG results ;
14. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyltransferase (GGT), total bilirubin (TBIL), blood creatinine (CRE), blood urea nitrogen (BUN), or international normalized ratio (INR) higher than the upper limit of normal (ULN) at screening, that are considered as clinically significant abnormalities by the investigator;
15. Part 2 only: abnormal sex hormone levels at screening that are considered clinically significant by the investigator;
16. Clinically significant abnormalities in thyroid function, parathyroid function, and neck ultrasound results at screening;
17. Women with positive pregnancy test result or those who are breastfeeding before dosing;
18. Positive hepatitis C virus antibody (HCV Ab), positive human immunodeficiency virus antibody (HIV Ab) or positive hepatitis B surface antigen (HbsAg) result at screening;
19. Unable to refrain from consuming grapefruit, pomelo, grapefruit juice, or pomelo juice from 48 hours prior to check-in until the end of the study;
20. Unable to refrain from consuming any foods or beverages containing caffeine or xanthine from 48 hours prior to check-in until the end of the study;
21. Unable to abstain from smoking/using tobacco products from 48 hours prior to check-in until the end of the study;
22. Unable to refrain from consuming alcohol from 48 hours prior to check-in until the end of the study;
23. Any history of narcotic use or drug abuse;
24. Any medical or other condition may affect the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Treatment -Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Day 4
  Number of participants with TEAEs and SAEs will be reported.
Part 2:Number of Participants With TEAEs and SAEs | Up to Day 12
  Number of female post-menopausal participants with TEAEs and SAEs will be reported.

SECONDARY OUTCOMES:
Parts 1 and 2: AUC0-t- Area Under the Drug Concentration-time Curve From Time 0 to the Last Sample Collection Time t for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  AUC0-t will be assessed and reported.
Parts 1 and 2: AUC0-infinity- Area Under the Drug Concentration-time Curve From 0 to Infinity for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  AUC0-infinity will be assessed and reported.
Parts 1 and 2: Cmax- Maximum Observed Plasma Concentration for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Cmax will be assessed and reported.
Parts 1 and 2: Tmax- Time to Reach the Maximum Plasma Concentration (Cmax) for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Tmax will be assessed and reported.
Parts 1 and 2: T1/2- Terminal Half-life for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  T1/2 will be assessed and reported.
Parts 1 and 2: CL/F- Apparent Clearance for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  CL/F will be assessed and reported.
Parts 1 and 2: Vd/F- Apparent Volume of Distribution for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Vd/F will be assessed and reported.
Part 2: Cmax,ss- Observed Maximum Concentration at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Cmax at steady state will be assessed and reported.
Part 2: Cmin,ss- Observed Minimum Concentration at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Cmin at steady state will be assessed and reported.
Part 2: Tmax,ss- Time of Cmax at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Tmax at steady state will be assessed and reported.
Part 2: Cavg,ss- Average Concentration at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Cavg at steady state will be assessed and reported.
Part 2: AUC0-τ- Area Under the Drug Concentration-time Curve During the Dosing Interval at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  AUC0-T at steady state will be assessed and reported.
Part 2: CLss/F- CL for Bioavailability at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  CL/F at steady state will be assessed and reported.
Part 2: T1/2,ss- Terminal Half-life at Steady State for GS1-144 | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  T1/2 at steady state will be assessed and reported.
Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose | Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Accumulation Ratio will be assessed and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia